CLINICAL TRIAL: NCT05413434
Title: The Effects of Exercise Training and Respiratory Muscle Training on Physical Fitness, Pulmonary Functions and METS Parameters in Individuals With METS
Brief Title: Exercise Training and Respiratory Muscle Training in Individuals With Metabolic Syndrome(METS)
Acronym: METS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hilal GÜNGÖR, Master off degree, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HacettepeKPR
Record Dates: First submitted 2022-03-06; First posted 2022-06-10 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; inspiratory muscle training; high intensity interval training; exercise
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Participant
Masking Description: The physician who referred patients to the study and the participants were blind to the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT with a supervisor (Experimental): These individuals will be given HIIT training on the treadmill, accompanied by a physiotherapist, 3 days a week for 8 weeks.
  Interventions: Other: exercise
- Hiit and respiratory muscle training with a supervisor (Experimental): HIIT program and respiratory muscle training will be applied to these individuals 3 days a week for 8 weeks.
  Interventions: Other: exercise; Device: inspiratory muscle training
- control group (No Intervention): The importance of physical activity will be explained and appropriate physical activity recommendations will be made.

INTERVENTIONS:
Other: exercise — high-intensity interval training will be performed on the treadmill.
  Arms: HIIT with a supervisor; Hiit and respiratory muscle training with a supervisor
Device: inspiratory muscle training — Respiratory muscle strength exercise will be performed with the respiratory muscle strengthening device 'POWERbreathe Classic Light Resistance'.
  Arms: Hiit and respiratory muscle training with a supervisor

SUMMARY:
The study will be conducted on individuals with Metabolic Syndrome. There are many studies showing that aerobic exercise provides significant improvements in waist circumference, fasting glucose, high-density lipoprotein cholesterol (HDL-C), Triglyceride (TG), systolic and diastolic blood pressure (SBP-DBP), and cardiorespiratory fitness on METS parameters. However, although the beneficial effects of physical activity are known, only half of the population adheres to the 150 minutes of moderate-intensity physical activity per week recommendation. High-intensity interval training (HIIT) is a type of training that uses near-maximal intensities in short-term sessions. HIIT has been used to improve compliance because it requires less time to treat patients with cardiometabolic disease. Compared to continuous aerobic exercise, this type of training has been shown to be an effective alternative for improving maximum oxygen consumption (VO2 max), blood pressure, heart function, glucose and lipid metabolism, and markers of oxidative stress and inflammation. In the literature, HIIT has been studied in patients with METS and has been shown to be effective. In addition, a study showed that seven-day respiratory muscle training was also effective on METS parameters, but there is no study showing the long-term effects of respiratory muscle training in this patient group. Therefore, in our study, researchers aimed to show the effects of respiratory muscle training given with HIIT on METS parameters.

DETAILED DESCRIPTION:
Metabolic syndrome (METS) is a systemic endocrinopathy characterized by the presence of risk factors such as abdominal obesity, glucose intolerance or diabetes mellitus, atherogenic dyslipidemia, hypertension, and a persistent proinflammatory profile. According to the International Diabetes Federation (IDF) definition of METS, almost 20-25% of the adult world population has METS, and people with METS are at risk of heart attack, stroke, type 2 diabetes (T2D), all-cause and cardiovascular death (approximately three times higher). In addition, modifiable risk factors such as physical inactivity, diet, and sedentary behavior have all been associated with increased prevalence of METS. Increasing incidence of METS, increase in morbidity and mortality necessitated the implementation of preventive strategies and the implementation of pharmacological and non-pharmacological treatments.

Studies in the literature have shown that vagal tone decreases and sympathetic tone increases in patients with METS. At the same time, impaired baroreflex sensitivity and decreased heart rate variability are observed in these patients. Changes in autonomic modulation cause the release of some bioactive molecules by affecting the endocrine and immune systems. In this case, increased sympathetic autonomic tone creates a cardiometabolic risk. In adults with METS, autonomic dysfunction appears to be more prominent in women than in men. Autonomic functions are impaired due to changes such as loss of lean body mass, increase in fat mass, increase in body mass, redistribution of fat from the periphery to the middle parts of the body, especially in postmenopausal women. As a result, increased blood pressure, impaired endothelial function, decreased glucose tolerance, and atherogenic changes in lipid and coagulation profiles can be observed. This increases the incidence of METS in postmenopausal women. Therefore, strategies to reduce the risk of metabolic syndrome have often been studied on women in the literature, and there is a need for studies involving men and new strategies.

Physical activity and exercise training are recommended as key prescriptions for the prevention and treatment of METS and low-grade chronic inflammation . Increase in physical exercise has been recommended for the prevention and primary treatment of cardiovascular disease (CVD) and METS because of the cardioprotective benefits associated with improved cardiorespiratory fitness (CRF). There are many studies showing that aerobic exercise provides significant improvements in waist circumference, fasting glucose, high-density lipoprotein cholesterol (HDL-C), TG, systolic and diastolic blood pressure (SBP-DBP), and cardiorespiratory fitness on METS parameters . However, although the beneficial effects of physical activity are known, only half of the population adheres to the 150 minutes of moderate-intensity physical activity per week recommendation. It has been shown that one of the main barriers to reaping health benefits and being more active is "lack of time". High-intensity interval training (HIIT) is a type of training that uses near-maximal intensities in short-term sessions. HIIT has been used to improve compliance because it requires less time to treat patients with cardiometabolic disease. Compared to continuous aerobic exercise, this type of training is an effective alternative to improve maximum oxygen consumption (VO2max), blood pressure, heart function, glucose and lipid metabolism, and markers of oxidative stress and inflammation . However, it has been seen that there are not enough studies on HIIT effectiveness on METS parameters in the literature. Therefore, researchers aimed to show the effects of HIIT training applied together with respiratory muscle training on METS parameters in patients with METS.

It has shown the beneficial effects of exercise training as well as inspiratory muscle training (IME) on autonomic function in patients with hypertension and heart disease . In a study, it was shown that 7-day inspiratory muscle training improved respiratory muscle functions and cardiac autonomic functions in postmenopausal women . As a result of this study, inspiratory muscle training has been proposed as a nonpharmacological strategy to improve autonomic modulation and reduce risk factors in individuals with METS, but further studies are required to confirm the long-term effects or effects of inspiratory muscle training in addition to classical exercise training protocols such as aerobic, resistance or combined training. are needed.

In a study conducted in healthy and middle-aged men and postmenopausal women in 2021, it was proven that high resistance inspiratory muscle strength training can improve blood pressure control and vascular endothelial function, and reduce the risk of cardiovascular disease and other clinical disorders. In this study, researchers presented the first evidence that inspiratory muscle strength training increases NO bioavailability, decreases systemic inflammation, and causes potentially beneficial changes in the plasma metabolome by increasing endothelial NO synthase activation and decreasing oxidative stress. In conclusion, it has been shown that inspiratory muscle strength training can be used as a promising lifestyle intervention to improve cardiovascular function and reduce the risk of other clinical disorders .

Since the long-term effects of respiratory muscle training in individuals with METS have not been examined in the literature; researchers planned this study to examine the effects of inspiratory muscle strength training added to aerobic exercise training (HIIT) on physical fitness, respiratory functions and METS parameters in individuals with METS.

ELIGIBILITY:
Inclusion Criteria:

* METS will be defined according to the National Adult Cholesterol Education Program Adult Treatment Panel III. Patients with at least three or more of the following five characteristics will be included in the study:
* Waist circumference ≥102 cm for men or ≥88 cm for women;
* blood pressure above 130/85 mmHg;
* Fasting blood glucose (FG) ≥100 mg/dL;
* Blood TG ≥150 mg/dL; and
* HDL-C < 40 mg/dL for men and < 50 mg/dL for women.
* Not participating in any physical activity program (≤2 physical activity days per week ≤ 30 minutes per session).
* 18 -65 years
* to walk and cooperate
* to participate in the research

Exclusion Criteria:

* heart failure,
* pectoris,
* of myocardial infarction or stroke in less than one year,
* hypertension,
* cardiovascular or kidney disease,
* with peripheral vascular disease and any disease associated with exercise intolerance will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
VO2max | 8 weeks
  Cardiorespiratory fitness will be performed using a cardiopulmonary exercise test (CPET) with a treadmill, using the measurement method (breath by breath) with each breath. The modified Bruce protocol will be applied.VO2max will be recorded in ml/kg/min.

SECONDARY OUTCOMES:
functional capacity | 8 weeks
  Functional capacity will be evaluated with a 1 minute sit-stand test. The number of sit-ups will be noted.
flexibility | 8 weeks
  flexibility will be evaluated with the functional reach test and sit and reach test. Results will be recorded in cm.
systolic and diastolic blood pressure | 8 weeks
  Systolic and diastolic blood pressure will be measured using a digital sphygmomanometer (BP710, Omron, Tokyo, Japan) and results will be recorded in millimeters of mercury (mmHg). After the participants rest for 5 minutes in a sitting position, two measurements will be taken with an interval of 1 minute. The average of the two measurements will be recorded in mmHg.
C-Reactive Protein (CRP) | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. CRP will be recorded in mg/dl.
Low Density Lipoprotein Cholesterol (LDL-C) | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. LDL-C will be recorded in mg/dl.
High Density Lipoprotein Cholesterol (HDL-C) | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. HDL-C will be recorded in mg/dl.
Total Cholesterol | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. Total Cholesterol will be recorded in mg/dl.
Triglycerides(TC) | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. TC will be recorded in mg/dl.
Fasting blood glucose | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. Fasting blood glucose will be recorded in mg/dl.
Hemoglobin A1c(HbA1c) | 8 weeks
  Fasting blood samples will be taken from the patients before and after the 8-week training, after 12 hours of fasting, at Hacettepe University Hospital, Department of Internal Medicine, General Internal Medicine. It will be held in the morning, 48 hours after the end of the training. HbA1c will be described in %.
spot urinalysis | 8 weeks
  In the urine analysis, albumin, protein and creatinine values will be recorded as mg/dl.
height | 8 weeks
  A non-flexible and sensitive up to 0.1 cm tape measure will be used to measure the height of the participants.Height will be recorded in centimeter(cm) .
body weight | 8 weeks
  Body Composition Scale will be used for body composition measurement . Body weight will be recorded in kilogram(kg).
Body mass index(BMI) | 8 weeks
  Weight and height will be combined to report BMI in kg/m^2.
Body fat ratio | 8 weeks
  Body fat ratio will be measured with 'MI Scala 2'. It will be recorded in %.
Respiratory function | 8 weeks
  Pulmonary function test parameters will be performed with a portable spirometer device in sitting position, taking into account the criteria of the American Thoracic Society and the European Respiratory Society. Forced Vital Capacity (FVC %), Forced expiratory volume (FEV1%) ,Peak expiratory flow (PEF %), forced mid-expiratory flow (FEF25-75%) will be recorded.
respiratory muscle strength | 8 weeks
  Respiratory muscle strength will be evaluated with a portable intraoral pressure gauge ('Micro Medical( MicroRPM), Rochester, UK). Maximal inspiratory pressure and maximal expiratory pressure values will be recorded in centimeters of water(cmH2O).

CONTACTS AND LOCATIONS:
Overall Officials: oğuz uyaroglu, PHD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol and data analysis will be shared with other researchers.